CLINICAL TRIAL: NCT01992172
Title: Pilot Study of Novel Topical Drug (Photocil) for the Treatment of Atopic Dermatitis
Brief Title: Photocil (Topical) for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Applied Biology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AB-DRUG-PHOTOCIL-AD-001
Record Dates: First submitted 2013-11-19; First posted 2013-11-25 (Estimated); Results first posted 2016-03-25 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Photocil for Atopic Dermatitis (Active Comparator): Active Drug - Photocil for Atopic Dermatitis
  Interventions: Drug: Photocil for Atopic Dermatitis
- Placebo - Sunscreen (SPF 2) (Placebo Comparator): Placebo - Sunscreen (SPF 2)
  Interventions: Other: Placebo - Sunscreen (SPF 2)

INTERVENTIONS:
Drug: Photocil for Atopic Dermatitis — Photocil for Atopic Dermatitis
  Other Names: Photocil for Atopic Dermatitis (U.S. FDA NDC: 54841-001-01)
  Arms: Photocil for Atopic Dermatitis
Other: Placebo - Sunscreen (SPF 2) — Placebo - Sunscreen (SPF 2)
  Arms: Placebo - Sunscreen (SPF 2)

SUMMARY:
Photocil is a topical drug (cream) that selectively delivers Narrow Band - Ultraviolet B (NB-UVB) therapy when exposed to sunlight. Photocil is intended to help protect users from non-therapeutic Ultraviolet B (UVB) radiation while selectively passing wavelengths of light in the NB-UVB range with peak transmission of 308nm. The aim of the study is to assess the safety and efficacy of Photocil in the treatment of atopic dermatitis.

DETAILED DESCRIPTION:
NB-UVB phototherapy is a common treatment for patients with atopic dermatitis, and has been reported to be safe and effective in numerous clinical trials. Clinical trials have reported achievement of Atopic Dermatitis Area Severity Index (ADASI)-75 in 50-70% of patients after 4-6 weeks of NB-UVB treatment.

Many drawbacks limit patients compliance, access, and acceptance of traditional NB-UVB phototherapy. The strict treatment regimen (2-3 sessions per week for an average of 12 weeks or more) performed at a specialized phototherapy clinic combined with high cost and low or no reimbursement make compliance and access a major drawback.

In order to address the drawbacks of phototherapy, we developed a novel topical cream - Photocil - that selectively delivers NB-UVB therapy when exposed to sunlight. When used with natural sunlight, Photocil provides a convenient alternative to traditional clinic based phototherapy; thus, has the potential to dramatically increase patient compliance and treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with atopic dermatitis confirmed by a dermatologist
* Atopic dermatitis lesions affecting at a minimum 5% of the facial, legs, or arms surface area
* Age: 18 to 65
* Participants able to give informed consent

Exclusion Criteria:

* Subject did not respond to prior phototherapy treatment
* Subject completed phototherapy for same lesion(s) in last 6 months
* Subject has previous history of skin cancer
* Subject has previous history of photosensitivity
* Subject has a history of herpes (HSV I or II) outbreaks
* Subject has previous history of autoimmune disease may be excluded at investigator's discretion
* Subject is currently taking of immunosuppressive or photosensitizing drugs
* Subject plans to use antibiotics, anti-fungal, calcineurin inhibitors or other drugs that may cause photosensitivity during the study period. These patients may be excluded at investigator's discretion
* Subject is pregnant or lactating women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-08; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John McCoy, PhD, Study Director — Applied Biology, Inc.
Locations (1):
- Physicians Institute, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Photocil for Atopic Dermatitis | Placebo - Sunscreen (SPF 2)
Started | 7 | 0
Completed | 7 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Photocil for Atopic Dermatitis | Placebo - Sunscreen (SPF 2) | Total
Number analyzed (Participants) | 7 | 0 | 7
Age, Categorical [Number; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 7 |  | 7
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (5.29) |  | 32.3 (5.29)
Gender [Number; unit: Participants]
  Female | 7 |  | 7
  Male | 0 |  | 0
Region of Enrollment [Number; unit: Participants]
  United States | 7 |  | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Pruritus Events in Last 30 Days
Time Frame: 30 days from baseline
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Photocil for Atopic Dermatitis | Placebo - Sunscreen (SPF 2)
Number analyzed (Participants) | 7 | 0
Events
  Baseline | 7.4 (2.9) |
  90 Day | 1.9 (1.5) |

ADVERSE EVENTS:
Arm/Group | Photocil for Atopic Dermatitis | Placebo - Sunscreen (SPF 2)
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/0
Other Adverse Events (participants affected / at risk) | 0/7 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days